CLINICAL TRIAL: NCT05245487
Title: Chemotherapy-induced Genomic Damage in Elderly Patients With Lymphoma: Prevalence, Evolution, and Clinical Consequences
Brief Title: Danish Elder Lymphoma Patient Hematopoietic Investigation
Acronym: DELPHI
Status: Recruiting | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Aalborg University Hospital (Other); Odense University Hospital (Other); Aarhus University Hospital (Other); Gødstrup Hospital (Other); Vejle Hospital (Other); Sonderborg Hospital (Other Government); Danish Cancer Society (Other); Zealand University Hospital (Other)
Responsible Party: Principal Investigator, Simon Husby, MD, PhD, MD, PhD, Rigshospitalet, Denmark
Other Study IDs: DELPHI
Record Dates: First submitted 2022-02-08; First posted 2022-02-18 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-04

CONDITIONS: Lymphoma; Chemotherapy-induced Neutropenia; Chemotherapy-Related Leukemia; Chemotherapeutic Toxicity
MeSH Terms: conditions — Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: DNA repair gene mutation analysis — Prospective monitoring of patients with next-generation sequencing for blood mutations

SUMMARY:
Every year approximately 300 Danish patients die from lymphoma. The median age at diagnosis is 70 years. Lymphoma can be efficiently treated with chemotherapy, and potentially cured. However, sufficient treatment is often hampered by toxicity, especially in elderly patients. It is also well known that the main risk factor for dying of lymphoma is age. New biologically targeted therapies with fewer side effects are becoming available for lymphoma treatment, however it is currently difficult to delineate which patients benefit from chemotherapy and which should be treated with novel expensive therapies.

Recently, it has been discovered that chemotherapy can provoke growth of patient blood cells with DNA mutations. This leads to increased rates of treatment side effects and excess mortality. These defects have so far only been examined in younger patients below 70 years of age, where they are found in roughly 10% of patients. It remains unknown to what extent elderly individuals are affected, but the investigators hypothesize that the proportion and negative effects are much larger.

Therefore, the investigators propose to investigate the frequency and evolution of these DNA mutations during chemotherapy in a prospective study of patients, who are either above 60 years of age and previously treated with chemotherapy for lymphoma in a nation-wide collaboration.

By using blood samples, advanced genetic analyses and patient-reported questionnaires, the investigators will study

* The prevalence of these mutations and their consequences for patient wellbeing, treatment side effects (such as anemia, infections etc.) and mortality
* The kinetics of these mutations during and after treatment, and explore possible evolutionary patterns of the inferred damages The investigators expect to include 300 patients in the study and that the first results will be ready in a timeframe of 4 years. The investigators hope to obtain new insights in the risk factors for physiological and mental health in lymphoma patients and thereby pave the way for improvements in wellbeing and survival of this underserved population.

DETAILED DESCRIPTION:
DELPHI is prospective nationwide observational study investigating blood mutations in patients with lymphoma.

Inclusion criteria:

* Diagnosis of B-cell Non-Hodgkin lymphoma
* In need of systemic treatment with second (2.) or higher line of active therapy for lymphoma
* 60 years of age or older (no age maximum)

Exclusion criteria:

* Unable to give written consent
* Non-Danish citizens

Patients will be included by their treating physcian at their local department. All analyses are centralized. Blood samples for research puporses will be taken before, midway (tipically before 3rd / 4th series depending on regimen) and 4-8 weeks after treatment. Also QOL questionaires will be sent electronically to the patients. The results of the tests performed will blinded to the patient and the treating physician.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of r/r B-cell Non-Hodgkin lymphoma
* In need of systemic treatment with second (2.) or higher line of active therapy for lymphoma
* 60 years of age or older (no age maximum)

Exclusion Criteria:

* Unable to give written consent
* Non-Danish citizens

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Danish citizens with r/r B-cell Non-Hodgkin lymphoma 60 years of age or older.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2035-01-01 (Estimated)

PRIMARY OUTCOMES:
Event-free survival (EFS) | 2 years
  EFS according to Revised Lugano Criteria

SECONDARY OUTCOMES:
Overall survival (OS) | 2 years
  OS

CONTACTS AND LOCATIONS:
Overall Officials: Simon Husby, MD PhD, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Dept. of Hematology, Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided